CLINICAL TRIAL: NCT03975231
Title: A Phase I Trial of Concurrent Intensity Modulated Radiation Therapy (IMRT) and Dabrafenib/Trametinib in BRAF Mutated Anaplastic Thyroid Cancer
Brief Title: Dabrafenib, Trametinib, and IMRT in Treating Patients With BRAF Mutated Anaplastic Thyroid Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21308; NCI-2019-02745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA246553 (NIH); OSU-17277 (Other: Ohio SU ID)
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: BRAF NP_004324.2:p.V600E; BRAF V600K Mutation Present; Thyroid Gland Anaplastic Carcinoma
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — dabrafenib; Radiotherapy, Intensity-Modulated; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dabrafenib, trametinib, IMRT) (Experimental): See Detailed Description
  Interventions: Drug: Dabrafenib; Radiation: Intensity-Modulated Radiation Therapy; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436A; GSK2118436
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This trial studies how well dabrafenib, trametinib, and intensity modulated radiation therapy (IMRT) work together in treating patients with BRAF mutated anaplastic thyroid cancer. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Giving dabrafenib, trametinib, and IMRT together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability (maximum tolerated dose [MTD]) of concurrent intensity modulated radiation therapy (IMRT) and BRAF-MEK inhibitors dabrafenib and trametinib in patients with BRAF-mutated anaplastic thyroid cancer.

SECONDARY OBJECTIVES:

I. To assess overall objective response rate, time to progression of local recurrence, progression free survival and overall survival.

II. To assess pharmacokinetics during concurrent IMRT and dabrafenib plus trametinib therapy.

III. To assess pharmacodynamics of dabrafenib plus trametinib induction therapy.

IV. To assess mechanism of resistance to dabrafenib plus trametinib and radiation therapy.

OUTLINE: This is a dose-escalation study of dabrafenib.

INDUCTION: Patients receive dabrafenib orally (PO) twice daily (BID) and trametinib PO once daily (QD) for 7-28 days in the absence of disease progression and unacceptable toxicity.

OPTIONAL SURGERY: Patients with resectable disease may undergo surgery 3 days after stop treatment of dabrafenib/trametinib, and move to Concurrent Radiation 14 days after surgery provided that surgical wound has healed. All other patients continue to receive dabrafenib PO BID and trametinib PO QD in the absence of disease progression and unacceptable toxicity.

CONCURRENT RADIATION: Patients receive dabrafenib PO BID and trametinib PO QD at weeks 6-7. Within 2.5 hours of morning doses of dabrafenib/trametinib administration, patients undergo intensity modulated radiation therapy (IMRT) on Monday-Friday delivered over 6.5 weeks in the absence of disease progression or unacceptable toxicity.

POST-RADIATION: Patients receive dabrafenib PO BID and trametinib PO QD for 4 weeks in the absence of disease progression and unacceptable toxicity.

MAINTENANCE: Patients with residual disease receive dabrafenib PO BID and trametinib PO QD in the absence of disease progression and unacceptable toxicity. Patients stop dabrafenib and trametinib 8 weeks after achieving complete response. Patients with no residual disease stop dabrafenib and trametinib, with the option of restarting dabrafenib and trametinib at time of disease recurrence.

After completion of study treatment, patients are followed up every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic (histologic or cytologic) diagnosis of anaplastic thyroid cancer (a diagnosis that is noted to be ?consistent with anaplastic thyroid cancer? with the presence of a thyroid mass is acceptable; pathology showing additional types of thyroid cancer is allowed)

  * Note: Tissue collection for central review is mandatory, but central review is not required for eligibility. Due to the aggressiveness of this disease, treatment will be started prior to central review.
* Presence of BRAF mutation (V600E or V600K) in tumor tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* Absolute neutrophil count > 1,000/mcL.
* Hemoglobin >= 9.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 9.0 g/dl is acceptable).
* Platelets > 75,000/mcL.
* Total bilirubin < 1.5 x institutional upper limit of normal (unless due to Gilbert?s disease).
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional upper limit of normal.
* Serum creatinine < 1.5 x institutional upper limit of normal.
* Female patients of childbearing potential are required to have a negative serum pregnancy test within 14 days prior to the first dose of study medication.
* Females are required to use an effective method of contraception from the time of negative serum pregnancy test, throughout the study duration, and for 4 months after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to study enrollment, for the duration of study participation, and for 16 weeks after completion of the last dose of study drug.
* Specific contraception requirements for females: Female subjects of childbearing potential must not become pregnant and are required to be sexually inactive by abstinence or use contraceptive methods with a failure rate of < 1%. Sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception. Contraceptive methods with a failure rate of < 1% include the following:

  * Intrauterine device (IUD) or intrauterine system (IUS) that meets the < 1% failure rate as stated in the product label,
  * Male partner sterilization (vasectomy with documentation of Azoospermia) prior to the female subject's entry into the study, and this male is patient?s sole sexual partner. For this definition, ?documented? refers to the outcome of the investigator's/qualified physician designee?s medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject?s medical records.
  * Double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam, gel, film, cream, suppository) These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring subjects understand how to properly use these methods of contraception.
* Specific contraception requirements for males: To prevent pregnancy in a female partner or to prevent exposure of any partner to the investigational product from a male subject?s semen, male subjects must use one of the following contraceptive methods during the study and for a total of 16 weeks following the last dose of study drug (based upon the lifecycle of sperm):

  * Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject for 14 days prior to first dose of study drug, through the dosing period, and for at least 16 weeks after the last dose of study drug. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Condom (during non-vaginal intercourse with any partner - male or female) OR
  * Condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository) (during sexual intercourse with a female).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with resectable stage IVA anaplastic thyroid cancer who are candidates for surgery and wish to proceed with surgery.
* Patients who have had external beam radiotherapy to neck or chest for cancer that would result in overlap of radiation therapy fields.
* Patients who have had cytotoxic chemotherapy, stereotactic brain radiation or external beam radiation within 2 weeks prior to study treatment initiation.
* Patients who have had oral multikinase inhibitors within 1 week prior to study treatment initiation.
* Patients that have not recovered from adverse events related to prior therapy for cancer to Common Terminology Criteria for Adverse Events (CTCAE) 4.03 grade 2 or less except for alopecia.
* Patients previously treated with potent BRAF inhibitor or MEK inhibitor. Previous treatment with sorafenib is permitted.
* Patients that are receiving any other investigational agent.
* Patients that are currently taking any prohibitive medication.
* Patients with a history of other active malignancy requiring cancer treatment.
* Patients with uncontrolled brain metastases. Patients who are on a stable dose of corticosteroids for more than 1 week or off corticosteroids for 2 weeks prior to study enrollment can be enrolled. Enzyme-inducing anti-epileptic drugs are not permitted.
* Patients with a known history of retinal vein occlusion (RVO), central serous retinopathy (CSR), uncontrolled glaucoma or ocular hypertension.
* Patients with class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Corrected QT (QTc) interval greater than or equal to 480 msecs (>= 500 msec for subjects with Bundle Branch Block).
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous (IV) antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and nursing women are excluded from this study because dabrafenib has the potential for teratogenic or abortifacient effects. In embroyfetal developmental studies in rats, developmental toxicities including reduced fetal body weight, embryo-lethality, cardiac ventricular septal defect malformations, delayed skeletal development and variation in thymic shape have been observed.
* Known human immunodeficiency virus (HIV)-positive patients or those on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of combination therapy of dabrafenib and trametinib administered concurrently with intensity-modulated radiation therapy (IMRT) | 1 year

SECONDARY OUTCOMES:
Objective response rate | 1 year
  Will be defined as the proportion of patients who have a partial response (PR), or complete response (CR) within the first 4 weeks of IMRT. Complete response (CR) and partial response (PR) will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be calculated with the exact binomial 95% confidence intervals.
Time to progression for local disease recurrence | 1 year
  Will be evaluated by RECIST criteria for disease limited to the radiation field (neck) following the first set of scans after completion of IMRT. Estimated by Kaplan-Meier method.
Overall survival | From the start date of the treatment to the date of death, assessed up to 1 year
  Estimated by Kaplan-Meier method.
Progression free survival | Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
  Estimated by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Sasan Fazeli, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Univ of Texas-M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu